CLINICAL TRIAL: NCT06057857
Title: An Experience of Oral Cancer Screening in Workplace: a Cross-sectional Study
Brief Title: Oral Cancer Screening in Workplace: a Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayat Gamal-AbdelNaser, Principle investigator, Cairo University
Other Study IDs: ACU-Med2
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Employees in Ahram Canadian university
  Interventions: Other: conventional oral examination

INTERVENTIONS:
Other: conventional oral examination — conventional oral examination

SUMMARY:
Employees are to be all screened for oral cancer in work place.

ELIGIBILITY:
Inclusion Criteria:

* adults

Exclusion Criteria:

* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all employees working in ACU
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Presence of lesion: oral cancer or oral potentially malignant lesions | upon study completion; an average of 3 months
  detected on examination

CONTACTS AND LOCATIONS:
Locations (1):
- Ahram Candian University, Giza, Egypt